CLINICAL TRIAL: NCT01512290
Title: Theta Burst Transcranial Magnetic Stimulation as Treatment for Auditory Verbal Hallucinations; a Placebo-controlled Trail
Brief Title: Theta Burst Transcranial Magnetic Stimulation as Treatment for Auditory Verbal Hallucinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Iris Sommer, Principle Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMCU_TBS
Record Dates: First submitted 2012-01-09; First posted 2012-01-19 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Auditory verbal hallucinations; Transcranial Magnetic stimulation; Theta Burst frequency
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theta burst treatment (Active Comparator): patients randomized to this arm will receive 10 TBS treatments distributed over 5 days
  Interventions: Other: Theta Burst Transcranial Magnetic Stimulation
- sham treatment (Placebo Comparator)
  Interventions: Other: Theta Burst Transcranial Magnetic Stimulation

INTERVENTIONS:
Other: Theta Burst Transcranial Magnetic Stimulation — This rTMS paradigm consists of 5 pulses at 50Hz repeated at 5Hz for 60 seconds with a total of 900 pulses per treatment

SUMMARY:
Auditory verbal hallucinations (AVH) are a characterising symptom of schizophrenia. In the majority of patients, these AVH respond well to antipsychotic medication. Yet, a significant minority continues to experience frequent AVH despite optimal pharmacotherapy. The number of alternative treatment options for this medication resistant group is currently low and most of them focus on coping with the hallucinations. Transcranial magnetic stimulation (TMS), in contrast, is a non-invasive technique of influencing cortical excitability. This technique has the potential to actually decrease the frequency and severity of medication resistant hallucinations.

Several previous studies have assessed efficacy of low frequency rTMS, with contradicting results. A previous large study by the investigators group could not demonstrate efficacy of low frequency rTMS. A new stimulation protocol using theta burst rTMS (TBS) could provide a more effective therapeutic option.

Objective: The present study aims to examine the efficacy of TBS on the severity of AVH. Study design: The objectives are tested in a randomized double blind placebo-controlled trail.

Study population: 60 patients with the diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder or psychosis not otherwise specified with frequent auditory verbal hallucinations will be included.

Intervention: The participant will receive either 10 TBS treatments or 10 placebo treatments consisting of 900 pulses each with a 30 minute interval on the left temporoparietal area, distributed over 5 treatment days. Stimulation will be at 80% of the motor threshold.

Main study parameters/endpoints: the main study parameter is the change in the severity of the AVH. The secondary study parameter is the number and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder or psychosis not otherwise specified.
* Age 18+ years.
* Frequent auditory verbal hallucinations (cut-off at >once an hour).
* Written informed consent.

Exclusion Criteria:

* Metal objects in or around the head that cannot be removed (i.e. cochlear implant, surgical clips, piercing, cardiac pacemaker, medicinal pumps)
* History of seizures
* Increased intracranial pressure due to infarcts or trauma.
* History of eye trauma with a metal object or professional metal workers
* Patients who are coercively treated at a psychiatric ward (based on a judicial ruling)
* Patients who are represented by a legal ward or under legal custody
* In female patients, there should be no possibility for pregnancy as determined with a pregnancy test
* Changes in the prescribed medication in a period of 2 weeks prior to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in severity and frequency of auditory verbal hallucinations | 1 week/ 1 month
  This is as experienced by the participant. The change in score on the Auditory Hallucination Assessment Scale (AHAS; Frederick, 2000), the PSYRATS (Haddock et al., 1999) and the total score on the PANSS item 3 (Kay et al. 1987), the item concerning the severity of the hallucinations, after one week of treatment end one month after treatment will be used for this outcome.

SECONDARY OUTCOMES:
Number and severity of adverse events | 1 week/ 1 month
  This is measured by the use of a selection of the Global index of Safety (Prieto, Sacristan & Gomez, 2004). The scores on this questionnaire are compared between the two conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Sommer, Prof., Dr., Study Director — UMC Utrecht; Anne Lotte Meijering, MSc., Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands